CLINICAL TRIAL: NCT03925246
Title: A Phase II Study From the POLA National Network of Nivolumab for Recurrent IDH Mutated High-Grade Gliomas
Brief Title: Efficacy of Nivolumab for Recurrent IDH Mutated High-Grade Gliomas
Acronym: REVOLUMAB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160923J; 2017-004140-38 (EudraCT Number)
Record Dates: First submitted 2019-03-14; First posted 2019-04-24 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: High Grade Glioma; Brain Cancer
Keywords: Recurrent high grade gliomas; IDH mutation; Immune Checkpoint inhibitor; Nivolumab
MeSH Terms: conditions — Glioma; Brain Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab is administered by a 30 minutes intravenous infusion at dose of 240 mg every 2 weeks for 8 doses (4 months), followed by a 60 minutes intravenous infusion at dose of 480 mg every 4 weeks for 8 doses (8 months) or until progression, death , unacceptable toxicity or end of the research.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab (Opdivo) is a potent human monoclonal antibody (mAb) of the IgG4 isotype designed to directly block the interaction between Programmed Cell Death 1 (PD-1) and its ligands, Programmed Death Ligand 1 (PD-L1) and PD-L2.
  Nivolumab is administered by a 30 minutes intravenous infusion at dose of 240 mg every 2 (+/- 2 days) weeks for 8 cycles (4 months), followed by a dose of 480 mg administered by a 60 minutes intravenous infusion every 4 weeks (+/-3 days) (beginning at cycle 9) for a total therapy duration of 1 year (maximum 16 cycles of treatment) or until progression, death, unacceptable toxicity.
  Other Names: Opdivo

SUMMARY:
Immune checkpoint blockade therapies targeting the immunomodulatory effect of cytotoxic T-lymphocyte antigen (CTLA-4) and programmed cell death-1/ Programmed death-ligand 1 (PD-1/PD-L1) have recently demonstrated survival benefit and durable response in phase III trials in several human cancers, especially in tumors that bear high mutation load and/or tumor-associated neoantigen signatures. The aim of these treatments is to restore effector T-cell function and antitumor activity, which could be enhanced in the context of high mutational/neoantigen load. In Isocitrate DeHydrogenase mutated High Grade Gliomas (IDHm HGGs), acquired resistance to alkylating chemotherapy frequently results from the inactivation of mismatch-repair (MMR) proteins which in turn leads to the acquisition of a hypermutator phenotype. These findings suggest that at least in a subset of recurrent IDHm HGGs immune checkpoint blockade therapies may be particularly effective. IDHm HGGs most frequently occur in young adults. The first line treatment consists of maximal safe surgical resection followed by radiotherapy and adjuvant alkylating chemotherapy (Temozolomide or Procarbazine-CCNU-Vincristine regimen (PCV)). Despite these treatments, most IDHm HGGs recurred in few years. There is no standard of care at recurrence and the median overall survival after it is less than 3 years.

The investigators make the hypothesis that treatment with the anti-PD-1 monoclonal antibody Nivolumab will improve 24 weeks progression-free survival in IDHm HGGs that have recurred after initial treatment with radiotherapy and alkylating chemotherapy.

DETAILED DESCRIPTION:
IDHm HGGs (High-Grade (grade III or IV) Gliomas that harbor mutations in Isocitrate Dehydrogenase 1 (IDH1) or Isocitrate Dehydrogenase 2 (IDH2)) most frequently occur in young adults. Favorable prognostic factors include high Karnofsky performance score, young age, 1p/19q codeletion and O6-methylguanine-DNA methyltransferase (MGMT) promoter methylation. Despite primary management, which consists of maximal safe surgical resection followed by radiotherapy and adjuvant alkylating chemotherapy with temozolomide (TMZ) or Procarbazine, CCNU, Vincristine (PCV), most IDHm HGGs recur, resulting in death with a median overall survival of 5 years. At recurrence, there is currently no standard of care. Because of the lack of clinical trials specifically designed for patients with relapsed IDHm HGGs, most patients receive alkylating chemotherapy (nitrosourea- or TMZ-containing regimens). However, these treatments have modest efficacy, as shown in several phase II trials that have reported response rates of 17-44% and 6-month progression-free survival (PFS6) of 29-51%. The efficacy of alkylating agents as DNA damaging agents is dependent on a functional MMR pathway. In IDHm HGGs, acquired resistance to alkylating chemotherapy can arise after the inactivation of MMR proteins, which in turn leads to the acquisition of a hypermutator phenotype. Paired analyses of newly diagnosed and recurrent tumors (after treatment with alkylating agents), have demonstrated that IDHm HGGs that recur after treatment with alkylating chemotherapy often harbor hypermutator phenotype associated with defects in the MMR pathway. While such MMR defects are extremely rare in newly diagnosed IDHm HGGs, MMR mutations were reported in 20-50% of patients with recurrent IDHm HGGs giving support that there is selective pressure to decreased MMR in glial tumors treated with alkylating chemotherapy. These findings suggest that, at least in a subset of recurrent IDHm HGGs, Nivolumab may be effective. Nivolumab has demonstrated overall survival (OS) benefit in multiple tumor types and has demonstrated a manageable safety profile in > 12300 subjects across all clinical trials. For monotherapy, the safety profile is similar across tumor types. Preliminary data from phase I and phase III trials in patient with gliomas have indicated that Nivolumab is well tolerated in patients with primary brain tumors. Yet, these tumors may represent particularly good candidates for immune checkpoint blockade therapies since they frequently develop a hypermutated phenotype after alkylating chemotherapy.

This is a phase II, open label, non-randomized multicentric trial evaluating the efficacy of Nivolumab in adults' patients with recurrent IDHm HGGs. The main objective is to evaluate the efficacy of Nivolumab, based on 24 weeks progression-free survival (PFS24w) rate as assessed by RANO criteria.

Nivolumab is administered by a 30 minutes intravenous infusion at dose of 240 mg every 2 (+/- 2 days) weeks for 8 cycles (4 months), followed by a dose of 480 mg administered by a 60 minutes intravenous infusion every 4 weeks (+/-3 days) (beginning at cycle 9) for a total therapy duration of 1 year (maximum 16 cycles of treatment) or until progression, death, unacceptable toxicity.

Patients will undergo efficacy assessments using magnetic resonance imaging (MRI) every 8 weeks (every 4 cycles during 8 first cycles, then every 2 cycles). Patient outcomes measures will be completed at the time of each imaging study. Toxicity assessments will occur before the initiation of each cycle. Health related Quality of life (EORTC QLQ-C30 and QLQ-BN20) will be assessed before day 1, every 4 cycles during 8 first cycles, then every 2 cycles.

* In case of discontinuation from study treatment for toxicity or severe adverse events, subject request or investigator decision :

  * PFS-24w assessment should be done at W24 +/- 2weeks if applicable
  * date of tumor progression according to RANO and iRANO criteria and date of death if applicable
* In case of end of treatment duration :

  * A brain MRI will be performed 4 weeks after the C16
  * After the end of the research, patient will be followed every 3 months as usual care, by phone, to record date of tumor progression according to RANO criteria and date of death, if applicable.
* Adverse events must be notified and documented by investigator for a minimum of 100 days after last dose of treatment. Drug-related toxicities should continue be followed until they resolve, return to baseline or are deemed irreversible.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of grade III or IV high-grade glioma
2. Tumor is mutated for IDH1 or IDH2 gene (detected by R132HIDH immunochemistry or IDH1/IDH2 sequencing)
3. Age between 18 and 85 years old
4. Recurrence after radiotherapy and at least one line of alkylating chemotherapy (Temozolomide or PCV (Procarbazine, CCNU, Vincristine) (Surgery at recurrence is allowed before trial inclusion)
5. Recurrence occurring more than 12 weeks from the end of the radiotherapy or occurring outside the irradiated volume
6. Karnofsky performance status > 50
7. Radiologically measurable disease based on RANO criteria. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
8. Patients must be able to taper steroids (preferably discontinued). Dose at inclusion must be ≤ 10 mg prednisone (or equivalent*). The decrease in dose will be evaluated by clinical examination, the ability to decrease the corticosteroids being related to the absence of increased headaches and the absence of increased of neurological disability (impaired alertness)
9. Available archived tissue for molecular (MGMT methylation, mutational load estimation) and immunohistochemical analysis (PD1, PD-L1, CD3, CD4, FoxP3, CD8, CD68, CD163, GFAP, olig2, ATRX, CIC, Ki67, P53)
10. The following laboratory values obtained ≤ 7 days prior to inclusion:

    * WBC ≥ 2000/μL
    * Neutrophils ≥ 1500/μL
    * Platelets ≥ 100 x103/μL
    * Hemoglobin > 9.0 g/dL
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

    Female CrCl = [(140 - age in years) x weight in kg x 1.04] / serum creatinine in µmol/l Male CrCl = ([140 - age in years) x weight in kg x 1.23] / serum creatinine in µmol/l
    * AST/ALT ≤ 3 x ULN
    * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)
    * Negative serum pregnancy test for women of childbearing potential
11. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 5 months after the last dose of study treatment (ie, 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo approximately five half-lives)
12. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment {i.e., 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo approximately five half-lives.}
13. Written informed consent dated and signed, prior to any study specific procedures (sampling, treatment and analyses).
14. Affiliation to a French social security system (recipient or assign) excluding AME.

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
3. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
4. Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol
5. Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity or congestive cardiac insufficiency
6. Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection, and/or detectable virus and a known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
7. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or > 1,5 mg dexamethasone or equivalent*) or other immunosuppressive medications within 14 days of first study treatment administration. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone or > 1,5 mg dexamethasone or equivalent, are permitted in the absence of active autoimmune disease.
8. Any chemotherapy, anticancer immunotherapy or anticancer agents within 4 weeks (6 weeks for nitrosourea) before the first dose of study treatment,
9. Receiving any other investigational agent or study drugs from a previous clinical study within 4 weeks before the first dose of study treatment (6 weeks for nitrosoureas).
10. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
11. History of allergy or Hypersensitivity to Nivolumab or to any of the excipients
12. Any unresolved toxicities (excepted alopecia), from prior therapy greater than CTCAE grade 1 at the time of inclusion.
13. Subjects with history of life-threatening toxicity, including hypersensitivity reaction, related to prior immunoglobulin treatment for another condition (except those considered unlikely to re-occur) or any other study drug component.
14. Surgical procedure < 7 days prior to first study treatment administration, vascular access device no restriction;
15. Subjects unable (e.g., due to pacemaker or ICD device) or unwilling to have a contrast-enhanced MRI of the head;
16. Known allergy or contraindication to Gadolinium;
17. Patients under guardianship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
24 weeks progression-free survival (PFS24w) rate, documented by RANO criteria | At 24 weeks (+/- 2 weeks) after treatment initiation
  Efficacy of Nivolumab will be based on PFS24w. PFS24w was defined by the percentage of patients alive without progression according to RANO criteria at 24 weeks +/- 2 weeks after treatment initiation.

SECONDARY OUTCOMES:
Progression-Free survival at 24 weeks (PFS24w) rate estimated by iRANO criteria | 24 weeks (+/- 2 weeks) after treatment initiation
  PFS24w was defined by the percentage of patients alive without progression according to iRANO criteria at 24 weeks +/- 2 weeks after treatment initiation.
Median progression-free survival (median-PFS) assessed by RANO criteria | From the date of treatment initiation until the date of first documented tumor progression or until the date of death due to any cause assessed up to 30 months
  Median-PFS is defined by the time in which fifty percent (50%) of patients have experienced tumor progression or death due to any cause. It will be documented using RANO criteria
Median progression-free survival (median-PFS) assessed by iRANO criteria | From the date of treatment initiation until the date of first documented tumor progression or until the date of death due to any cause assessed up to 30 months
  Median-PFS is defined by the time in which fifty percent (50%) of patients have experienced tumor progression or death due to any cause. It will be documented using iRANO criteria
Overall survival (OS) | From the date of the treatment initiation until the date of death due to any cause, assessed up to 30 months
  Overall survival is defined as the time from treatment initiation to death due to any cause
Overall response rate (ORR) assessed by RANO criteria | From the date of the treatment initiation to the date of the end of treatment, assessed up to 30 months
  Overall response rate is defined by the percentage of patients with at least a complete response and partial response using RANO criteria documented during treatment
Overall response rate (ORR) assessed by iRANO criteria | From the date of the treatment initiation to the date of the end of treatment, assessed up to 30 months
  Overall response rate is defined by the percentage of patients with at least a complete response and partial response using iRANO criteria documented during treatment
Duration of response assessed by RANO criteria | From the date of the treatment initiation until the date of tumor progression, assessed up to 30 months
  Duration of response is defined by the time from confirmation of stable, partial and complete response using RANO criteria until the tumor progression has been shown
Duration of response assessed by iRANO criteria | From the date of the treatment initiation until the date of tumor progression, assessed up to 30 months
  Duration of response is defined by the time from confirmation of stable, partial and complete response using iRANO criteria until the tumor progression has been shown
Longitudinal changes in quality of life (EORTC QLQ-C30 and BN20) | Before day 1 (t0) then every 4 cycles during 8 first cycles, then every 2 cycles until cycle 16 (1 cycle = 28 days)
  Data at each time point will be compared to t0 (before first infusion of Nivolumab)
Safety: Type, frequency and severity of adverse events and serious adverse events | Up to 30 months after the date of the treatment initiation
  The adverse events will be described and graded according to the revised NCI Common Terminology Criteria V4.03 for Adverse Events (CTCAE V4.03)

CONTACTS AND LOCATIONS:
Overall Officials: DEHAIS Caroline, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (7):
- France (7):
  - Groupe Hospitalier Saint-André, Bordeaux
  - Hospices Civils de Lyon, Hôpital Pierre Wertheimer, Bron
  - AP-HM, La Timone, Hôpital Universitaire, Marseille
  - Institut de Cancérologie de l'Ouest (ICO) - site CLCC René Gauducheau, Nantes
  - AP-HP - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - AP-HP - Hôpital Saint-Louis, Paris
  - IUCT Oncopole - CLCC Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Result] Picca A, Touat M, Belin L, Gourmelon C, Harlay V, Cuzzubbo S, Cohen-Jonathan Moyal E, Bronnimann C, Di Stefano AL, Laurent I, Lerond J, Carpentier C, Bielle F, Ducray F, Dehais C; POLA Network. REVOLUMAB: A phase II trial of nivolumab in recurrent IDH mutant high-grade gliomas. Eur J Cancer. 2024 May;202:114034. doi: 10.1016/j.ejca.2024.114034. Epub 2024 Mar 22. PMID 38537315